CLINICAL TRIAL: NCT01437839
Title: An Open Label, Randomized, 2-period Crossover Study Evaluating Single Dose Food Effect On Apixaban Commercial Image Tablets In Healthy Subjects
Brief Title: Food Effect Study For Apixaban Commercial Image Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B0661019
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Food effect study; Pharmacokinetics; Apixaban
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Period I: fasting state, Period II: fed state
  Interventions: Drug: Apixaban
- 2 (Experimental): Period I: fed state, Period II: fasting state
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Period I: 1 x 5 mg Commercial Image Tablet in fasting state(single dose on Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period), Period II: 1 x 5 mg Commercial Image Tablet in fed state (single dose on Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period)
  Arms: 1
Drug: Apixaban — Period I: 1 x 5 mg Commercial Image Tablet in fed state(single dose on Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period), Period II: 1 x 5 mg Commercial Image Tablet in fasting state (single dose on Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period)
  Arms: 2

SUMMARY:
To evaluate the effect of food on the pharmacokinetics of apixaban administered as commercial image tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* History or evidence of abnormal bleeding or coagulation disorder (eg, easy bruising or gingival bleeding, prolonged bleeding after dental extraction, postpartum, or after trauma, wounds or surgery) and/or having a first degree relative under 50 years of age with a history of abnormal bleeding or coagulation disorder

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cmax | dosing to 3 days
AUC(INF) | dosing to 3 days

SECONDARY OUTCOMES:
AUC(tlqc) | dosing to 3 days
Tmax | dosing to 3 days
t1/2 | dosing to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- [Derived] Song Y, Chang M, Suzuki A, Frost RJ, Kelly A, LaCreta F, Frost C. Evaluation of Crushed Tablet for Oral Administration and the Effect of Food on Apixaban Pharmacokinetics in Healthy Adults. Clin Ther. 2016 Jul;38(7):1674-1685.e1. doi: 10.1016/j.clinthera.2016.05.004. Epub 2016 Jun 10. PMID 27292282
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0661019&StudyName=Food%20Effect%20Study%20For%20Apixaban%20Commercial%20Image%20Tablets